CLINICAL TRIAL: NCT00071357
Title: Use of Dynamic Contrast-Enhanced Magnetic Resonance Imaging to Assess Tumor-Associated Vasculature in Patients With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040003; 04-N-0003
Record Dates: First submitted 2003-10-20; First posted 2003-10-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Breast Neoplasms
Keywords: Microarray; Herceptin; Trastuzumab; Carcinoma; Proteomics; Breast Cancer; Metastatic Breast Cancer; Metastatic Breast Tumor
MeSH Terms: conditions — Breast Neoplasms; Carcinoma

SUMMARY:
This study will examine a non-invasive method to assess vasculature, that is, the development of a blood supply necessary to the growth of tumors. The hope is to identify the way that genes are expressed within the tumor itself, from areas shown as low flow versus those shown as high flow on dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI).

Most patients with solid epithelial cancers, those that develop on free surfaces or linings inside the body, die because of the distant spread of tumors-metastasis. After that spread, a cure is more difficult than if the tumors were detected early or locally. Tumors develop a new supply of blood. Traditional anticancer therapies have had the goal of causing a decline in the tumor. Yet by focusing on the tumor's blood supply, microscopic differences between tumors and clonal differences within tumors may be avoided. Doing so may overcome tumor resistance to treatment and may result in treatments that can be more universally applied across tumor types.

Female patients 18 years of age enrolled in the protocol Analysis of Brain Metastasis in Patients with Breast Cancer, with and without Over-Expression of HER-2, who will undergo an MRI scan immediately before surgery will be invited to participate in this study. Patients seen in the oncology outpatient clinic of the NIH Clinical Center or by referral from outside physicians may be eligible for this study.

Participants will undergo DCE-MRI immediately before the craniotomy-the surgery scheduled-in conjunction with other clinically indicated MRI. The preoperative MRI will take about 30 minutes, and the DCE-MRI will take no more than 15 minutes. During the MRI, patients will lie still on a table that can slide in and out of a metal cylinder surrounded by a strong magnetic field. They may be asked to lie still for up to 5 minutes at a time. As the scanner takes pictures, there will be loud knocking noises, and the patients will wear earplugs to muffle the sound. Patients will be able to communicate with the MRI staff at all times during the scan and may ask to be moved out of the machine at any time. During part of the MRI, patients will receive a contrast agent, one that is gadolinium-based, into a vein. This agent changes the relative brightness or contrast on the MRI image under some conditions. Before that agent is used, patients will be asked about any previous allergic reactions to gadolinium-based contrast agents.

DETAILED DESCRIPTION:
Introduction: Metastasis of epithelial tumors, such as breast cancer, to the brain is a common problem, with significant consequences with respect to neurological dysfunction and shortening of survival. One necessary step for tumor growth anywhere is the development of a blood supply.

Objectives: We seek to compare a new, non-invasive method of assessing neo-vascularization, dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) with a gold-standard-microvessel counts-and to see if we can identify gene expression patterns within the tumor itself, from areas shown as low flow versus those that are high-flow on DCE-MRI if there are features within the tumor itself that influence the degree of neovascularization. This prospective study will only be utilized in conjunction the protocol entitled "Analysis of Brain Metastasis in Patients with Breast Cancer, with and without over-expression of HER-2" that is evaluating breast tumors metastatic to the brain.

Study Population: A series of women with breast cancer metastatic to the brain who do (n=39) or do not (n=39) over-express the growth factor receptor, HER-2, entered into a prospective trial in which pre-operative MRI imaging is performed as a matter of standard medical practice. At the time of this pre-operative MR, we propose to add one additional, 10-minute MR series, a dynamic, contrast-enhance image to assess the extent of blood flow through various aspects of the tumor.

Anticipated Risks and Benefits: There are no obvious risks or benefits to patients who participate in this protocol. It is felt that this study involves no more than minimal risk.

Estimation of Outcome/Potential Meaning: We believe that this protocol will help us identify tumors with higher or lower degrees of neovascularization as well as identify tumor-intrinsic factors via microarrays performed on microdissected tissues. This is becoming an important issues as cytostatic treatments, such as anti-angiogenic agents, enter the clinical area, and are used singly or in combination with cytotoxic therapies.

ELIGIBILITY:
Inclusion Criteria:

1. A woman with a known or with radiographic evidence of a breast neoplasm metastatic to the brain, who has agreed to participate in the protocol "Analysis of Brain Metastasis in Patients with Breast Cancer, with and without over-expression of HER-2," and who will undergo a pre-operative MR scan immediately before surgery.
2. Medically-indicated (diagnostic and/or therapeutic) brain tumor resection.
3. Informed consent from female patient, age 18 or older. In general, patients less than 18 years of age rarely have breast cancer metastatic to the brain.

Exclusion Criteria:

1. Inability to provide informed consent prior to surgery.
2. Medical conditions that cannot be corrected prior to surgery that would be standard contraindications for craniotomy (brain tumor patients).
3. Conditions that preclude MR imaging of the brain (Patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices) or known allergy to gadolinium.
4. Men

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78
Dates: Start 2003-10; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Steeg PS. Metastasis suppressors alter the signal transduction of cancer cells. Nat Rev Cancer. 2003 Jan;3(1):55-63. doi: 10.1038/nrc967. PMID 12509767
- [Background] Chambers AF, Groom AC, MacDonald IC. Dissemination and growth of cancer cells in metastatic sites. Nat Rev Cancer. 2002 Aug;2(8):563-72. doi: 10.1038/nrc865. PMID 12154349
- [Background] Patchell RA, Tibbs PA, Walsh JW, Dempsey RJ, Maruyama Y, Kryscio RJ, Markesbery WR, Macdonald JS, Young B. A randomized trial of surgery in the treatment of single metastases to the brain. N Engl J Med. 1990 Feb 22;322(8):494-500. doi: 10.1056/NEJM199002223220802. PMID 2405271